CLINICAL TRIAL: NCT02420496
Title: Enteral Fish Oil is Superior to Ursodeoxycholic Acid (UDCA) and Placebo (?) for the Treatment of Cholestasis in Infants
Brief Title: Enteral Fish Oil is Superior to Ursodeoxycholic Acid (UDCA) and Placebo for the Treatment of Cholestasis in Infants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20150165H
Record Dates: First submitted 2015-04-01; First posted 2015-04-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Cholestasis; Liver Disease
Keywords: Parental nutrition; associated
MeSH Terms: conditions — Cholestasis; Liver Diseases | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enteral fish oil (Experimental): Infants will receive enteral fish oil at a dose of 1mg/kg/day divided in two daily doses given enterally.
  Interventions: Drug: Enteral fish oil
- UDCA (ursodeoxycholic acid) (Active Comparator): Infants will receive UDCA at a dose of 10mg/kg/dose in two daily doses given enterally
  Interventions: Drug: Ursodeoxycholic Acid
- Placebo (Placebo Comparator): Infant will receive placebo in two daily doses given enterally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enteral fish oil
  Other Names: Nordic Natural Omega 3
  Arms: Enteral fish oil
Drug: Ursodeoxycholic Acid
  Other Names: Actigall
  Arms: UDCA (ursodeoxycholic acid)
Drug: Placebo
  Other Names: Sterile Water
  Arms: Placebo

SUMMARY:
To investigate the effect of enteral fish oil and UDCA on the time of cholestasis resolution and other markers of parenteral nutrition-associated liver disease.

ELIGIBILITY:
Inclusion Criteria:

Neonates admitted to the Neonatal Intensive Care Unit (NICU) at University Hospital (UH) in San Antonio, Texas, who:

1. Are >14 days old and <24 months of age
2. Have a serum direct bilirubin of ≥2 mg/dL
3. Are receiving <3 g/k/day of Intralipid via TPN
4. Are expected to remain hospitalized for at least an additional 21 days

Exclusion Criteria:

1. Have a congenitally lethal condition (e.g. Trisomy 13)
2. Have clinically severe bleeding not able to be managed with routine measures
3. Have evidence of a viral hepatitis or primary liver disease as the etiology of their cholestasis
4. Have other health problems such that survival is extremely unlikely even if cholestasis improves
5. Known allergy to eggs or fish products
6. Receiving IV Fish oil
7. Phenobarbital therapy at enrollment

Ages: 14 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Direct Bilirubin | Evaluated every 7 days up to 180 days
  Direct bilirubin less than 1 mg/dL considered resolution of cholestasis

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Blanco, M.D., Principal Investigator — University of Texas
Locations (1):
- University Hospital, San Antonio, Texas, United States

REFERENCES:
- [Background] Kelly DA. Liver complications of pediatric parenteral nutrition--epidemiology. Nutrition. 1998 Jan;14(1):153-7. doi: 10.1016/s0899-9007(97)00232-3. PMID 9437702
- [Background] Christensen RD, Henry E, Wiedmeier SE, Burnett J, Lambert DK. Identifying patients, on the first day of life, at high-risk of developing parenteral nutrition-associated liver disease. J Perinatol. 2007 May;27(5):284-90. doi: 10.1038/sj.jp.7211686. Epub 2007 Mar 8. PMID 17344923
- [Background] Nathan JD, Rudolph JA, Kocoshis SA, Alonso MH, Ryckman FC, Tiao GM. Isolated liver and multivisceral transplantation for total parenteral nutrition-related end-stage liver disease. J Pediatr Surg. 2007 Jan;42(1):143-7. doi: 10.1016/j.jpedsurg.2006.09.049. PMID 17208555
- [Background] Colomb V, Jobert-Giraud A, Lacaille F, Goulet O, Fournet JC, Ricour C. Role of lipid emulsions in cholestasis associated with long-term parenteral nutrition in children. JPEN J Parenter Enteral Nutr. 2000 Nov-Dec;24(6):345-50. doi: 10.1177/0148607100024006345. PMID 11071594
- [Background] Javid PJ, Greene AK, Garza J, Gura K, Alwayn IP, Voss S, Nose V, Satchi-Fainaro R, Zausche B, Mulkern RV, Jaksic T, Bistrian B, Folkman J, Puder M. The route of lipid administration affects parenteral nutrition-induced hepatic steatosis in a mouse model. J Pediatr Surg. 2005 Sep;40(9):1446-53. doi: 10.1016/j.jpedsurg.2005.05.045. PMID 16150347
- [Background] Calder PC. Use of fish oil in parenteral nutrition: Rationale and reality. Proc Nutr Soc. 2006 Aug;65(3):264-77. doi: 10.1079/pns2006500. PMID 16923311
- [Background] Clayton PT, Whitfield P, Iyer K. The role of phytosterols in the pathogenesis of liver complications of pediatric parenteral nutrition. Nutrition. 1998 Jan;14(1):158-64. doi: 10.1016/s0899-9007(97)00233-5. PMID 9437703
- [Background] Alwayn IP, Andersson C, Zauscher B, Gura K, Nose V, Puder M. Omega-3 fatty acids improve hepatic steatosis in a murine model: potential implications for the marginal steatotic liver donor. Transplantation. 2005 Mar 15;79(5):606-8. doi: 10.1097/01.tp.0000150023.86487.44. PMID 15753852
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Premkumar MH, Carter BA, Hawthorne KM, King K, Abrams SA. Fish oil-based lipid emulsions in the treatment of parenteral nutrition-associated liver disease: an ongoing positive experience. Adv Nutr. 2014 Jan 1;5(1):65-70. doi: 10.3945/an.113.004671. PMID 24425724
- [Background] Chen CY, Tsao PN, Chen HL, Chou HC, Hsieh WS, Chang MH. Ursodeoxycholic acid (UDCA) therapy in very-low-birth-weight infants with parenteral nutrition-associated cholestasis. J Pediatr. 2004 Sep;145(3):317-21. doi: 10.1016/j.jpeds.2004.05.038. PMID 15343182
- [Background] Thibault M, McMahon J, Faubert G, Charbonneau J, Malo J, Ferreira E, Mohamed I. Parenteral nutrition-associated liver disease: a retrospective study of ursodeoxycholic Acid use in neonates. J Pediatr Pharmacol Ther. 2014 Jan;19(1):42-8. doi: 10.5863/1551-6776-19.1.42. PMID 24782691
- [Background] Tillman EM, Crill CM, Black DD, Hak EB, Lazar LF, Christensen ML, Huang EY, Helms RA. Enteral fish oil for treatment of parenteral nutrition-associated liver disease in six infants with short-bowel syndrome. Pharmacotherapy. 2011 May;31(5):503-9. doi: 10.1592/phco.31.5.503. PMID 21923431
- [Background] Yang Q, Ayers K, Welch CD, O'Shea TM. Randomized controlled trial of early enteral fat supplement and fish oil to promote intestinal adaptation in premature infants with an enterostomy. J Pediatr. 2014 Aug;165(2):274-279.e1. doi: 10.1016/j.jpeds.2014.02.002. Epub 2014 Mar 12. PMID 24630347